CLINICAL TRIAL: NCT02986815
Title: [11C]Acetate PET in Patients With Glioma
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: low enrollment
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STU 052016-034
Record Dates: First submitted 2016-11-22; First posted 2016-12-08 (Estimated); Last update posted 2021-03-25 (Actual); Status verified 2021-03

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- [11C]Acetate Brain Imaging (Experimental): [11C]Acetate will be administered The patient will have one intravenous line placed prior to [11C]Acetate administration. The patient will receive the low-dose CT portion of a PET/CT scan, after which [11C]Acetate will be administered intravenously over approximately 1 min at a dose of 0.3 mCi/kg (maximum 30 mCi) and followed by a saline flush. The injection and imaging procedure will be terminated in any patient who exhibits anaphylaxis, significant dyspnea or chest pain. The administering physician will stay with the patient for at least 15 min after injection and will remain in the Clinical PET Facility through the duration of the imaging procedure.
  Interventions: Other: [11C]Acetate Brain Imaging

INTERVENTIONS:
Other: [11C]Acetate Brain Imaging — Patients will be imaged on a Siemens Biograph 64 slice PET CT scanner. After placing the patient on the scanner and securing the head in a head restraint, a low dose CT of the brain will be acquired. Images with 3 mm slice thickness and spaced at 1.5 mm intervals will be reconstructed in a 300 mm field of view. The purpose of the CT is for image localization and attenuation correction and it is not considered to be a diagnostic quality CT. Following the completion of the CT, the [11C]Acetate will be administered. A dynamic PET image will be acquired in 3D list mode for a total of 30 minutes.

SUMMARY:
At each point that the patient will have [11C]-Acetate PET study, this will be compared with standard clinical MR imaging. Abbreviations: XRT - radiation therapy; TMZ - temozolomide (chemotherapy)

Quantitative Image Data Analysis: The [11C]-Acetate uptake in tumor sites from images will be analyzed qualitatively by visual assessment, quantitatively using a standard uptake value (SUV) in the tumor relative to the contralateral normal brain, and the parameters obtained by compartmental modeling of dynamic data.

DETAILED DESCRIPTION:
1. [11C]Acetate Administration [11C]Acetate will be administered in the Clinical PET Facility located on the 2nd floor of the Clements Imaging Building at UT Southwestern. Upon arrival, the patient will have an opportunity to have questions answered regarding the procedure. The patient will have one intravenous line placed prior to [11C]Acetate administration. The patient will receive the low-dose CT portion of a PET/CT scan, after which [11C]Acetate will be administered intravenously over approximately 1 min at a dose of 0.3 mCi/kg (maximum 30 mCi) and followed by a saline flush. The injection and imaging procedure will be terminated in any patient who exhibits anaphylaxis, significant dyspnea or chest pain. The administering physician will stay with the patient for at least 15 min after injection and will remain in the Clinical PET Facility through the duration of the imaging procedure. All adverse events occurring post [11C]Acetate infusion will be recorded within a 24-hour period. The adverse events to be specifically monitored during the infusion include localized discomfort at the IV injection site, pain, respiratory difficulties, flushing, dizziness, pruritus/rash, and any other symptoms that could be secondary to an anaphylactic reaction. The subject will be instructed to report any subjective symptoms or sensory changes noted.

Patients will be imaged on a Siemens Biograph 64 slice PET CT scanner. After placing the patient on the scanner and securing the head in a head restraint, a low dose CT of the brain will be acquired. Images with 3 mm slice thickness and spaced at 1.5 mm intervals will be reconstructed in a 300 mm field of view. The purpose of the CT is for image localization and attenuation correction and it is not considered to be a diagnostic quality CT. Following the completion of the CT, the [11C]Acetate will be administered as described in Section VI.F.3.b.

A dynamic PET image will be acquired in 3D list mode for a total of 30 minutes. From the list mode data a flow image series will be constructed as follows:

* 12 frames x 10 seconds each (out to 2 minutes post-injection)
* then 6 frames x 30 seconds each
* then 1 frame x 60 seconds each

A second series will be -reconstructed to demonstrate dynamic brain regional metabolism as follows:

* 12 frames x 10 seconds each (out to 2 minutes post-injection)
* then 8 frames x 30 seconds each (from 2 to 6 minutes)
* then 4 frames x 60 seconds each (from 6 to 10 minutes)
* then 2 frames of 300 seconds each (from 10 to 20 minutes)
* then 1 frame of 600 seconds (from 20 to 30 minutes) Reconstructions will be performed with a 128 x 128 image matrix using 3D OSEM (4 iterations, 21 subsets) and a 3 mm Gaussian filter.

  3. Study Procedures and Schedule of Events:
  1. Initial visits prior to [11C]Acetate PET/CT:

     Patients who are identified as potential candidates for the study will be approached to explain the study and to obtain their written informed consent to be enrolled in the protocol. The following additional patient data will be obtained: histologic diagnosis (if a surgical procedure has been carried out), IDH mutational status, age at radiologic diagnosis, weight, full medical and neurological history and physical exam. Correlative imaging will be performed using MR brain, with and without gadolinium, within 14 days prior to enrollment. In addition, when available, 2-hydroxyglutarate (2HG) MR spectroscopy will be available for review and determination of 2HG concentration. For patients referred from outside UTSW and Parkland hospital, patient records and imaging will be reviewed to determine eligibility for the study and to obtain baseline comparative imaging scans.
  2. Day of baseline and follow up [11C]Acetate scans:

     [11C]Acetate PET/CT scan performed at baseline and at the time of clinical follow up; 3 months for grade 2 glioma patients on standard follow up, 2-3 months after treatment for patients being imaged pre- and post-treatment. The patient will be positioned supine in the PET/CT scanner for a dynamic scan over the brain. Patients will have two intravenous lines placed, one in each arm. [11C]Acetate PET/CT will be performed using the standard dose of 0.3 mCi/kg up to a maximum of 30mCi for [11C]Acetate. A single imaging field over the brain will be imaged dynamically for 30 min following the start of a 1-min intravenous infusion of [11C]Acetate, as described in Section VI.F.2.

     4. General Concomitant Medication and Supportive Care Guidelines Any adverse effects, related or non-related to the injection of [11C]Acetate, will be treated as clinically indicated with no study-related restrictions.

     5. Duration of Therapy and Follow-up: This is an observational study and patients will remain on study for the duration of their clinical follow up, as determined by their treating physician. [11C]Acetate PET scan timing will be determined based on their individual clinical course.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 18 and older, of any ethnic group
* Spanish-speaking patients will be eligible
* Histological diagnosis of glioma or
* Brain MR imaging suggestive of a glioma or 2HG > 2mM by MR spectroscopy in patients who have not had a surgical procedure to establish the diagnosis.
* Karnofsky Performance status > 70%
* Negative serum pregnancy test or child bearing potential terminated by surgery, radiation, menopause or current use of two approved methods of birth control
* Patient able and willing to provide informed consent

Exclusion Criteria:

* Patient or legal parent/guardian unable to provide informed consent
* Psychiatric or addictive disorders that preclude obtaining informed consent
* Karnofsky Performance status < 70%
* NYHA class III and IV congestive heart failure
* Unstable angina
* Pregnant or lactating women
* Women of childbearing potential who refuse a pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2017-01-24 (Actual); Primary Completion 2020-05-05 (Actual); Study Completion 2020-05-05 (Actual)

PRIMARY OUTCOMES:
Visual differences from normal brain in patients with grades 2, 3 or 4 gliomas | Every 3 months for 24 months
  Visual assessment and SUV with standard clinical MR imaging assessment.using T2/FLAIR and gadolinium enhancement.

SECONDARY OUTCOMES:
Decrease in [11C]Acetate uptake following treatment of grade 2 glioma | Every 3 months for 24 months
  Change from baseline in single imaging field over the brain, imaged dynamically for 30 minutes following the start of a 1-min intravenous infusion of [11C]Acetate
Decrease in [11C]-acetate uptake following treatment of grade 3 and 4 glioma | Every 3 months for 24 months
  Change from baseline in single imaging field over the brain, imaged dynamically for 30 minutes following the start of a 1-min intravenous infusion of [11C]Acetate.
Change in [11C]-acetate uptake following treatment at time of progression in grade 3 and 4 gliomas | Every 3 months for 24 months
  Change from baseline in single imaging field over the brain, imaged dynamically for 30 minutes following the start of a 1-min intravenous infusion of [11C]Acetate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No